CLINICAL TRIAL: NCT04050475
Title: A Randomized-controlled Pilot Study to Evaluate the Efficacy of a Fasting Mimicking Diet Added to Functional Therapy for Depression
Brief Title: The Evaluation of the Efficacy of a Fasting Mimicking Diet Added to Functional Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Collaborators: University of Palermo (Other); Centro Studi Psicoterapia Neo-Funzionale (Unknown)
Responsible Party: Principal Investigator, Giuseppe Maniaci, Principal Investigator, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AOPalermo
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: Depression; Fasting Mimicking Diet; Functional Therapy; Lifestyle Medicine; Health Psychology; Psychosomatic
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: After a psychiatric, psychological and anthropometric assessment, depressed patients were randomly assigned to psychotherapy and diet (PSY-FMD) or only psychotherapy (PSY) groups. PSY-FMD participants received 20 individual sessions of Functional Psychotherapy. Each session attended twice a week for the first 8 weeks and once a week for the remaining 4. Furthermore, they received a nutritional consultation and prescription of a Fasting Mimicking Diet. PSY group received just the psychotherapy protocol and the nutritionist prescribed to keep a food diary without changing their habitual diet style. All patients were retested at the end of the treatment (3 months later) and at follow-up 3 months after the last session.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients were advised that they would have received a psychological treatment and a nutritional consultation in order to evaluate the possibility of the prescription of a diet, investigating on their diet habits The investigator wasn't informed about the randomization procedures of the two groups.
  A clinical psychologist administered the psychological tests separately in the same treatment centre were the patients received the protocol and he wasn't aware about the randomization arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSY-FMD (Experimental): Subjects randomized in the PSY-FMD group carried out the Functional Therapy protocol over 20 individual sessions, which were scheduled twice a week for the first two months and once a week for the last month (three months total). The treatment program was specifically manualized for treating depression with the aim to increase mood, self-esteem and quality of life. Furthermore, patients followed a Fasting Mimicking Diet (FMD) protocol consisting of 3 cycles of 5 days a month each: the first day of the diet provided 1090 kcal (10% protein, 56% fat, 34% carbohydrate), the days 2-5 were identical in the formulation and provided 725 kcal (9-10% protein, 44-56% fat, 34-47% carbohydrate). Between cycles of FMD the subjects stuck to a free diet. At the end of the treatment all patients were re-tested through the same assessment protocol and the same things was realized at the follow-up (three months later the end of the treatment).
  Interventions: Dietary Supplement: Fasting Mimicking Diet
- PSY (No Intervention): Subjects randomized into the control group (PSY) completed the same Functional Therapy program without practicing any diet. Specifically, at the end of the nutritional consultation the nutritionist suggested them to keep a food diary without changing their habitual diet style.

INTERVENTIONS:
Dietary Supplement: Fasting Mimicking Diet — The Fasting Mimicking Diet is a low-calorie, five-day eating program meant to promote weight loss and provide the same benefits as more traditional fasting methods.
  Arms: PSY-FMD

SUMMARY:
Depression has to be considered as a systematic illness involving the whole body, it is often associated with low-grade inflammation and alterations of the microbiome. In this regard, an unhealthy diet increases the risk of the onset of this disorder, therefore an integrated treatment including a healthy diet could be more effective. The aim of our study were to verify the efficacy of a structured FT program, delivered in individual setting, for patients with depression (PSY group), and to verify whether the association of a FMD protocol with the structured FT program significantly improves clinical outcomes (PSY-FMD group). After a psychiatric, psychological and anthropometric assessment, depressed patients were randomly assigned to psychotherapy and diet (PSY-FMD) or just psychotherapy (PSY). PSY-FMD participants received 20 individual sessions of Functional Psychotherapy. Each session attended twice a week for the first 8 weeks and once a week for the remaining 4. Furthermore, they received a nutritional consultation and prescription of a Fasting Mimicking Diet. PSY group received just the psychotherapy protocol and the nutritional consultation. All patients were retested at the end of the treatment and at follow-up 3 months after the last session. In both groups was highlighted a strong effectiveness of treatments on depression, self-esteem and quality of life. In the PSY-FMD group compared to PSY a significant effect was found on the improvement of self-esteem and quality of life. Furthermore, a significant reduction of BMI was found in the PSY-FMD group. The current study supports the effectiveness of the combination of psychotherapy with a fasting mimicking diet in adult depressed patients.

DETAILED DESCRIPTION:
Depression is considered as a systemic illness affecting the whole body and increasing the risk of several diseases. Several studies showed an important link between depression and inflammation. Indeed, depression is associated with the activation of peripheral and central immune-inflammatory pathways indicated by increased levels of proinflammatory cytokines, such as Interleukin-1 β (IL-1β), Interleukin-6 (IL-6), Tumor necrosis factor-α (TNFα) and Interferon-γ (IFNγ). Furthermore, depressed patients present high levels of C-reactive Protein (CRP).

Furthermore, several studies underlined the existence of a link between depression and alterations of the microbiome, as the gut microbiota is implicated as an important health determinant relevant to mental health Several psychotherapy programs have demonstrated to be effective in treating depression, such as Cognitive-Behavioral Therapy (CBT), psychodynamic approaches and mind-body approaches, such as yoga and meditation.

There is some empirical evidence suggesting that the Functional Therapy (FT) approach, that represents an integrated body-mind therapy, highlights the possibility of inducing real changes of the cognitive, emotional and psychological systems through direct body intervention. The purpose of FT for depression is to increase mood and self-esteem through several bodily, cognitive, and emotional techniques by helping depressed patients to improve the Basic Experiences of the Self (BES) altered in this disorder. Furthermore, the integrated treatment provides an overall framework to facilitate lifestyle changes reinforcing assertiveness and self-efficacy.

A considerable body of literature highlighted the role of a healthy diet for reducing the risk of depression. On the other side, a diet based on Western dietary pattern is associated with depressed mood and anxiety. The typology of diet also modulates several key biological processes that underscore mood disorders, such as brain plasticity, stress response system, inflammation, and oxidative processes. Furthermore, practicing a Western dietary pattern implicates a negative effect on our immune system, associating with higher inflammation, and food-related inflammation is associated to increased risk of depression. Indeed, high stress levels and poor diet may lead to a disruption of the Hypothalamic-Pituitary-Adrenal (HPA) axis, with consequent increasing of cortisol's level, low-grade systemic inflammation and oxidative stress.

In this regard, a specific typology of diet oriented on fasting has proved to be effective on several parameters related to health. Cheng and colleagues (2014) found that periodic prolonged fasting promote stress resistance, self-renewal, and lineage-balanced regeneration; moreover, their results showed that cycles of fasting reduced the immunosuppression and mortality caused by chemotherapy in mice. A gradual calorie restriction, mimicking fasting effects but providing all macro- and micro-nutrients on mice rejuvenated the immune system, extended longevity, bring to lowered visceral fat, reduced cancer incidence and retarded bone mineral density loss. Furthermore, the authors found that in old mice FMD cycles promoted hippocampal neurogenesis and improved cognitive performance and motor coordination. Moreover, a Fasting Mimicking Diet protocol was associated with a significant reduction of TNFα, IL-1β and IL-6, and this decrease could positively influence the mood.

Given these premises, the aim of this clinical trial were:

1. Verify the efficacy of a structured FT program, delivered in individual setting, for patients with depression (PSY group);
2. Verify whether the association of a FMD protocol with the structured FT program significantly improves clinical outcomes (PSY-FMD group).

Patients were enrolled from January 2018 to March 2019 and were recruited via advertisement posted in our outpatient clinic. For the recruitment a structured telephone screening helped the researchers to investigate on some exclusion criteria. Then a consultation with a clinical psychologist and with a psychiatrist were programmed together with the administration of the psychological tests. Psychological assessment included an ad-hoc sociodemographic questionnaire; a shortened version of Wechsler Adult Intelligence Scale - Revised (WAIS-R); Millon Clinical Multiaxial Inventory-III (MCMI-III); Beck Depression Inventory-II (BDI-II); Basic Self-Esteem Scale (Basic SE); World Health Organization Quality of Life-BREF (WHOQOL-BREF). Anthropometric parameters included weight, height and waist circumference.

Six different therapists with a 4-year postgraduate training on FT applied the intervention. All therapists took part to a refresher training oriented to the application of the structured FT protocol for depression. Each therapist treated four patients. A nutritionist prescribed the FMD protocol after a consultation. After the assessment, eligible subjects were randomized in the PSY-FMD group or in the PSY group and were assigned to the next therapist on a time capacity list. A block randomization was used, so that number of patients per condition were balanced within therapists. The resulting samples comprised 20 depressed subjects. Four patients dropped out. There were no pre-treatment group differences on age, sex, marital status and years of education. Furthermore, both groups were homogeneous on Intelligence Quotient, the presence of psychiatric comorbidities or personality disorders, as well as for the level of depression, self-esteem, quality of life and BMI.

Ten subjects were randomized in the PSY-FMD group and they carried out the FT protocol over 20 individual sessions, which were scheduled twice a week for the first two months and once a week for the last month (three months total). None of the patients were undergoing psychopharmacological treatment. The treatment program was specifically manualized for treating depression with the aim to increase mood, self-esteem and quality of life. Specifically, the treatment program was oriented towards the reduction and/or elimination of mood unbalance through several bodily, cognitive and emotional techniques, such as deep breathing, specific guided imagery, techniques for improving assertiveness and for improving social abilities. Furthermore, patients recruited in the PSY-FMD group, followed a FMD protocol consisting of 3 cycles of 5 days a month each: the first day of the diet provided 1090 kcal (10% protein, 56% fat, 34% carbohydrate), the days 2-5 were identical in the formulation and provided 725 kcal (9-10% protein, 44-56% fat, 34-47% carbohydrate). Between cycles of FMD the subjects stuck to a free diet.

Ten subjects were randomized into the control group (PSY) and completed the same FT program without practicing any diet. Specifically, at the end of the nutritional consultation the nutritionist suggested them to keep a food diary without changing their habitual diet style.

At the end of the treatment all patients were re-tested through the same assessment protocol (psychological tests, anthropometric measures and nutritional consultation) to analyse the achievement of the expected outcomes and the same things was realized at the follow-up (three months later the end of the treatment).

Group differences in demographic features and pre-treatment measures were analysed with independent samples t-tests and χ2- tests. In order to evaluate the pre-post treatment alterations, a repeated ANOVA measurement was used at baseline, at the end of treatment and at the follow-up period. All analyses assumed an alpha risk of 5%. All statistical analyses were conducted using Statistical Package for Social Science for Windows 22.0.

ELIGIBILITY:
Inclusion Criteria:

* a score at the Beck Depression Inventory - II (BDI-II) over than 13 at the time of initial assessment;
* age from 18 to 60 years old;
* seeking treatment for mood problems;
* not involved in a concurrent treatment;
* without any psychopharmacological treatment for depression in the previous 12 months;
* without any practice of yoga or meditation;

Exclusion Criteria:

* a current or lifetime diagnosis of psychotic disorders, borderline, schizotypal, or antisocial personality disorder, active suicidal ideation with a plan, eating disorders, bipolar disorder, primary anxiety disorder
* a past or present of drug abuse or drug addiction (excluding nicotine)
* chronic inflammation diseases
* eating disorders
* IQ less than 65
* BMI less than 18.5 or more than 30
* severe hepatic failure
* serious infections (such as HIV, hepatitis B and C)
* cancer in the previous 6 months
* regular use of anti-inflammatory drugs for more than 15 days/month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
severity of depressive symptoms measured by the second version of the Beck-Depression-Inventory (BDI-II) | end of the treatment (three months) and three months later (follow-up)
  change of depression symptoms (measured through Beck Depression Inventory -II). Total score from 0 to 63. Higher values represent worst depression symptoms

SECONDARY OUTCOMES:
self-esteem measured by the Basic Self-Esteem Scale | end of the treatment (three months) and three months later (follow-up)
  change of self-esteem (measured through Basic Self-Esteem Scale). Percentiles scores were used (from 0 to 100). Higher values indicate a better self-esteem
quality of life measured by the WHO Quality of Life-BREF (WHOQOL-BREF) | end of the treatment (three months) and three months later (follow-up)
  change of Quality of Life (measured through World Health Organization Quality of Life BREF). Subscales: physical health, psychological health, social relationships, and environment. Score from 0 to 100. Higher values represent a better quality of life in each area

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Psychiatry, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maniaci G, La Cascia C, Giammanco A, Ferraro L, Chianetta R, Di Peri R, Sardella Z, Citarrella R, Mannella Y, Larcan S, Montana S, Mirisola MG, Longo V, Rizzo M, La Barbera D. Efficacy of a fasting-mimicking diet in functional therapy for depression: A randomised controlled pilot trial. J Clin Psychol. 2020 Oct;76(10):1807-1817. doi: 10.1002/jclp.22971. Epub 2020 May 11. PMID 32394438